CLINICAL TRIAL: NCT01240928
Title: A Phase Ib Trial of MK-2206 (an AKT Inhibitor) in Combination With Endocrine Therapy in Patients With Hormone Receptor-Positive Breast Cancer
Brief Title: MK-2206+Endocrine Therapy in Patients With Hormone Receptor-Positive Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding not available, study did not open to accrual and will not open in future
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Vandana Abramson, Assistant Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 1029
Record Dates: First submitted 2010-10-26; First posted 2010-11-15 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-2206 + exemestane +/- goserelin (Experimental): Oral MK-2206 and oral exemestane and subcutaneous goserelin (for pre-menopausal participants only)
  Interventions: Drug: MSK-2206; Drug: Exemestane; Drug: Goserelin

INTERVENTIONS:
Drug: MSK-2206 — Level 1: MK-2206 135mg weekly
Drug: Exemestane — Level 1: Exemestane - 25mg daily
Drug: Goserelin — Level 1: Goserelin- 3.6mg monthly for pre-menopausal subjects only

SUMMARY:
This is a phase Ib trial that evaluates the safety and tolerability of MK-2206 given in combination with exemestane +/- goserelin in pre- and post-menopausal patients with hormone receptor-positive metastatic breast cancer.

DETAILED DESCRIPTION:
The phase II portion of this trial will be listed under a separate NCT number.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stage IV invasive mammary carcinoma, documented by histological analysis, ER-positive and/or PR-positive by immunohistochemistry (IHC), previous endocrine therapy in the metastatic setting or had metastatic recurrence within 6 months of adjuvant endocrine therapy. May have measurable or non-measurable disease, both are allowed. Any number of prior hormone or chemotherapy agents are acceptable
2. Female and ≥ 18 years of age on the day of signing informed consent
3. Performance status of 0 or 1 on the ECOG Performance Scale
4. Adequate organ function as indicated by the following laboratory values:

   Hematological:
   * Absolute neutrophil count (ANC) ≥ 1,500 /μL
   * Platelets ≥ 100,000 /μL
   * Hemoglobin ≥ 9 g/dL

   Renal:

   -Serum creatinine or calculated creatinine clearance† - ≤ 1.5 x upper limit of normal (ULN) OR ≥60 mL/min for patients with creatinine levels > 1.5 x institutional ULN

   Hepatic:
   * Serum total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN or ≤5 x ULN in patients with known liver metastasis

   Coagulation:
   * Prothrombin time (PT)/INR ≤ 1.2 x ULN
   * Partial thromboplastin time (PTT) ≤ 1.2 x ULN

   Metabolic:

   -HBA1C ≤ 8%

   † Creatinine clearance calculated per institutional standard

   ‡ Fasting defined as at least 8 hours without oral intake
5. Female patient of childbearing potential must have negative serum or urine pregnancy test β-hCG within 72 hours prior to receiving the first dose of study medication
6. Post-menopausal female subjects defined prior to protocol enrollment by any of the following:

   * At least 55 years of age
   * Under 55 years of age and amenorrheic for at least 12 months or follicle-stimulating hormone (FSH) values ≥ 40 IU/L and estradiol levels < or equal to 20IU/L
   * Prior bilateral oophorectomy or prior radiation castration with amenorrhea for at least 6 months
7. Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent
8. Able to swallow capsules and has no surgical or anatomical condition that will preclude swallowing and absorbing oral medications on an ongoing basis
9. May receive concurrent radiation therapy to painful bone metastases or areas of impending bone fracture as long as radiation therapy is initiated prior to study entry. Those who have received prior radiotherapy must have recovered from any toxicity induced by this treatment (toxicity grade ≤ 1)

Exclusion Criteria:

1. Chemotherapy, radiotherapy, or biological therapy within 3 weeks (6 weeks for nitrosoureas, mitomycin C or bevacizumab), or not recovered from the adverse events due to previous agents administered more than 4 weeks prior to Study Day 1. If residual toxicity from prior treatment,toxicity must be ≤ Grade 1
2. Must be at least 4 weeks post-major surgical procedure, and all surgical wounds must be fully healed
3. Currently participating or has participated in a study with an investigational compound or device within 30 days of Study Day 1
4. Known active CNS metastases and/or carcinomatous meningitis. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 1 month prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis (2)off steroids used to minimize surrounding brain edema
5. Primary central nervous system tumor
6. Known hypersensitivity to the components of study drug or its analogs
7. History or current evidence of clinically significant heart disease including:

   * congestive heart failure, unstable angina pectoris,
   * cardiac arrhythmia,
   * history or current evidence of a myocardial infarction during the last 6 months,and/or a current ECG tracing that is abnormal in the opinion of the treating Investigator,
   * baseline QTc prolongation > 450 msec (Bazett's Formula). Medications included in Arizona CERT Lists 1 and 2 (Appendix D) must be excluded. The concomitant use of drugs that are associated with increased risk for QT prolongation should be avoided in patients with congenital long QT syndrome (Appendix D, Arizona CERT List 3). Similarly, the concomitant use of drugs that are weakly associated with QT prolongation should be generally avoided (Appendix D, Arizona CERT List 4). Arizona CERT List 3 and 4 drugs should be used at the discretion of the Investigator and restricted where applicable. Any therapy given with these drugs should be used with caution, and patients receiving these medications should be carefully monitored.
8. Evidence of clinically significant bradycardia (HR <50), or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree AV block (Mobitz Type 2), or patients taking beta blockers, non-dihydropyridine calcium channel blockers, or digoxin
9. Uncontrolled hypertension (i.e., 160/90 mHg SiBP). Patients who are controlled on antihypertensive medication will be allowed to enter the study
10. At significant risk for hypokalemia (e.g., patients on high dose diuretics, or with recurrent diarrhea)
11. Poorly controlled diabetes defined as HbA1C > 8%
12. History or current evidence of any condition, therapy, or lab abnormality that might confound the study results, interfere with the patient's participation for the full study duration, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
13. Known psychiatric or substance abuse disorders that would interfere with cooperation with trial requirements
14. Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse
15. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
16. Human Immunodeficiency Virus (HIV)-positive
17. Known history of Hepatitis B or C or active Hepatitis A
18. Symptomatic ascites or pleural effusion. Patient who is clinically stable following treatment for these conditions is eligible
19. Receiving treatment with oral corticosteroids (note: inhaled corticosteroids are permitted)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Tolerability of MK-2206 given in combination with exemestane +/- goserelin, as measured by maximum tolerated dose (MTD). | at 4 weeks
  The MTD will be defined as the highest dose tested in which a dose-limiting toxicity is experienced by 0 out of 3 or 1 out of 6 patients among the dose levels.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety of MK-2206 when combined with exemestane +/- goserelin | At 4 weeks
  Number of participants with worst-grade toxicity at each of five grades following NCI Common Toxicity Criteria: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, disabling, 5 = death
Characterize the effect of MK-2206 in combination with exemestane +/- goserelin based on PI3K, AKT, and PTEN mutations, as measured by immunohistochemistry and the SNaPshot assay. | After collection of tumor tissue
  Using tumor blocks from previous surgeries or fresh biopsies of accessible metastatic sites

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Abramson, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center